CLINICAL TRIAL: NCT06183645
Title: ActiCIDP : Exploratory Study on the Feasibility of Predicting CIDP Patients' Evolution Decline During Intravenous Immunoglobulins Treatment Adaptation.
Brief Title: Exploratory Study on Predicting CIDP Patients' Decline During IV Immunoglobulin Treatment Adaptation Feasibility.
Acronym: ActiCIDP
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: SYSNAV (Industry); Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Stéphanie DELSTANCHE, Coordinator of reference center for neuromuscular diseases, Centre Hospitalier Universitaire de Liege
Other Study IDs: ActiCIDP
Record Dates: First submitted 2023-12-14; First posted 2023-12-27 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Actimyo; Accelerometry; Daily living
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Actimyo — Participants will wear 2 Actimyos in everyday life. Actimyo is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.

SUMMARY:
ActiCIDP is a monocentric academic study. Patients with Chronic inflammatory demyelinating polyradiculoneuritis may be included on a voluntary basis.

The investigators plan to include a group of approximately 40 patients with CIDP.

The investigators have planned to assess patient every three months for a year. After each visit, participants will wear Actimyo for one month daily.

DETAILED DESCRIPTION:
On each visit, participants will undergo a clinical examination with MRC sum score, a mISS score and a I-RODS score.

They will perform few tests 6-minutes walk test (6MWT), a myogrip measurement, and a 9 Hole Peg Test (9HPT) and will answer to some questionaires (mISS, INCAT and PGIC).

Actimyo is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CIDP or possible CIDP based on 2021 EAN/PNS criteria2.
* Treated with IVIg (≤1g/kg/3-8week)
* Clinically Stable disease for 3 months (according to treating physician opinion).
* No treatment withdrawal failure within 1 year
* Age over 18 years

Exclusion Criteria:

* Significant cognitive or communication disorders
* Surgery or serious traumatic injury ≤ 6 months
* Non ambulant patient
* Current participation to a therapeutic trial
* Anti-myeline antibodies (anti-MAG) positive or nodo-paranodopathy
* Other autoimmune disease that requires Corticosteroids, IVIg, Plasma Exchange treatment
* Pregnancy or breastfeeding
* Any other condition that, according to the investigator, could significantly interfere with patient evaluation or safety.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with Chronic inflammatory demyelinating polyradiculoneuritis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
95th centile of stride velocity | 1 year
  95th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo) in real-life (meter per second).
50th centile of stride velocity | 1 year
  50th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo) in real-life (meter per second).
95th centile of stride length | 1 year
  95th centile of stride length obtained with a magneto-inertial sensor (Actimyo) in real-life (meter).
50th centile of stride length | 1 year
  50th centile of stride length obtained with a magneto-inertial sensor (Actimyo) in real-life (meter).

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Poleur, Dr, Principal Investigator — CHR Citadelle
Locations (1):
- CHR Citadelle, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No